CLINICAL TRIAL: NCT06085534
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficiency and Safety of LNK01001 Capsule in Patients With Ankylosing Spondylitis
Brief Title: A Study of LNK01001 Capsule in Patients With Ankylosing Spondylitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lynk Pharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LK001203
Record Dates: First submitted 2023-10-10; First posted 2023-10-17 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LNK01001 Dose A (Experimental): Participants were randomized to receive LNK01001 capsule dose A BID orally for 12 weeks in Period 1. At Week 13, participants were re-randomized to LNK01001 dose A or B capsule BID orally for 12 weeks in Period 2.
  Interventions: Drug: LNK01001
- LNK01001 Dose B (Experimental): Participants were randomized to receive LNK01001 capsule dose B BID orally for 12 weeks in Period 1. At Week 13, participants were re-randomized to LNK01001 capsule dose A or B BID orally for 12 weeks in Period 2.
  Interventions: Drug: LNK01001
- placebo (Placebo Comparator): Participants were randomized to receive a placebo capsule twice a day (BID) orally for 12 weeks in Period 1. At Week 13 participants were re-randomized to receive LNK01001 capsule dose A or B BID orally for 12 weeks in Period 2.
  Interventions: Drug: LNK01001; Drug: Placebo

INTERVENTIONS:
Drug: LNK01001 — Capsules for oral use
Drug: Placebo — Capsules for oral use
  Arms: placebo

SUMMARY:
The objective of this study was to evaluate the safety and efficacy of multiple doses of LNK01001 monotherapy versus placebo in the treatment of adults with active Ankylosing Spondylitis

DETAILED DESCRIPTION:
This study includes two periods. In Period 1, Participants who meet eligibility criteria will be randomized in a 1:1:1 ratio to receive a twice daily oral LNK01001 Dose A or LNK01001 Dose B or a matching placebo for 12 weeks. Participants who receive a placebo in Period 1 will be re-randomized at Week 13 in a 1:1 ratio to receive a twice daily oral LNK01001 Dose A or LNK01001 Dose B for 12 weeks (period 2). Those participants, based on the ASAS40 response, who receive LNK01001 (Dose A or Dose B) in Period 1 may switch to receive a different treatment dose for 12 weeks (period 2).

ELIGIBILITY:
Inclusion Criteria:

* Participants between ≥ 18 and ≤75 years of age.
* Diagnosis of ankylosing spondylitis (AS) who meet the 1984 revised New York Criteria for AS.
* Subjects must have disease activity at Screening and baseline visit.
* Subjects have received NSAIDs treatment but still have active AS, or subjects have an intolerance to or contraindication for NSAIDs.
* Never received tumor necrosis factor alpha (TNFα) treatment or prior exposure to ≤1 before randomization.

Exclusion Criteria:

* History of infection or any active infection.
* History of malignancy or current diagnosis of malignancy within 5 years before screening visit.
* Previous recipient of an organ transplant.
* Diagnosis of active uveitis within 6 months before randomization.
* Subject with any major surgery (including joint surgery) within 3 months before randomization or planned major surgery within the first 6 months during study.
* Prior exposure to Janus Kinase (JAK) inhibitor.
* Subjects who are allergy to any component of the study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving 40% Improvement in ASAS Score at Week 12. | Week 12
  ASAS40 response was defined as improvement of ≥ 40% relative to Baseline and absolute improvement of ≥ 2 units (on a scale from 0 to 10) in ≥ 3 of the following 4 domains with no deterioration (defined as a net worsening of > 0 units) in the potential remaining domain:
  Patient's global assessment of disease activity, measured on a numeric rating scale (NRS) from 0 (no activity) to 10 (severe activity); Pain, measured by the total back pain NRS from 0 (no pain) to 10 (most severe pain); Function, measured by the Bath Ankylosing Spondylitis Functional Index (BASFI) which consists of 10 items assessing participants' ability to perform activities on an NRS ranging from 0 (easy) to 10 (impossible); Inflammation, measured by the mean of the 2 morning stiffness-related Bath AS Disease Activity Index (BASDAI) NRS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each on a scale from 0 (none/0 hours) to 10 (very severe/2 hours or more duration).

SECONDARY OUTCOMES:
Percentage of Participants Achieving 40% Improvement in ASAS Score at Week 8,16,24 | Week 8,16,24
  ASAS40 response was defined as improvement of ≥ 40% relative to Baseline and absolute improvement of ≥ 2 units (on a scale from 0 to 10) in ≥ 3 of the following 4 domains with no deterioration (defined as a net worsening of > 0 units) in the potential remaining domain:
  Patient's global assessment of disease activity, measured on a numeric rating scale (NRS) from 0 (no activity) to 10 (severe activity); Pain, measured by the total back pain NRS from 0 (no pain) to 10 (most severe pain); Function, measured by the Bath Ankylosing Spondylitis Functional Index (BASFI) which consists of 10 items assessing participants' ability to perform activities on an NRS ranging from 0 (easy) to 10 (impossible); Inflammation, measured by the mean of the 2 morning stiffness-related Bath AS Disease Activity Index (BASDAI) NRS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each on a scale from 0 (none/0 hours) to 10 (very severe/2 hours or more duration).
Percentage of Participants Achieving 20% Improvement in ASAS Score. | Week 8,12,16,24
  ASAS20 response was defined as an improvement of ≥ 20% and an absolute improvement of ≥ 1 unit (on a scale of 0 to 10) from Baseline in at least 3 of the following 4 domains, with no deterioration (defined as a worsening of ≥ 20% and a net worsening of ≥ 1 units [on a scale of 0 to 10]) in the remaining domain:
  Patient's global assessment of disease activity, measured on a NRS from 0 (no activity) to 10 (severe activity); Pain, measured by the total back pain NRS from 0 (no pain) to 10 (most severe pain); Function, measured by the BASFI which consists of 10 items assessing participants' ability to perform activities on an NRS ranging from 0 (easy) to 10 (impossible); Inflammation, measured by the mean of the 2 morning stiffness-related BASDAI NRS scores (items 5 [level of stiffness] and 6 [duration of stiffness]) each on a scale from 0 (none/0 hours) to 10 (very severe/2 hours or more duration).
Percentage of Participants with an ASAS 5/6 response. | Week 8,12,16,24
  ASAS5/6 consists of 6 domains: the 4 used in ASAS20 (Patient's Global Assessment of Disease Activity, spinal pain, function, inflammation plus spinal mobility and an acute phase reactant, C Reactive Protein (CRP). ASAS 5/6 is defined as ≥20% improvement in at least 5 domains and no worsening in the remaining domain.
Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | Week 8,12,16,24
  The BASDAI assesses disease activity by asking the participant to answer 6 questions (each on an 11 point numeric rating scale [NRS]) pertaining to symptoms experienced for the past week. For Questions 1 to 5 (level of fatigue/tiredness, level of AS neck, back or hip pain, level of pain/swelling in joints, other than neck, back or hips, level of discomfort from any areas tender to touch or pressure, and level of morning stiffness), the response is from 0 (none) to 10 (very severe); for Question 6 (duration of morning stiffness), the response is from 0 (0 hours) to 10 (≥ 2 hours). The overall BASDAI score ranges from 0 to 10. Lower scores indicate less disease activity.
Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) | Week 8,12,16,24
  The Bath Ankylosing Spondylitis Functional Index is a validated index to determine the degree of functional limitation in patients with AS. BASFI consists of 10 questions assessing participants' ability to perform activities such as putting on socks, bending, reaching, getting up from the floor or an armless chair, standing, climbing and other physical activities. Each item is scored on a NRS ranging from 0 (easy to perform an activity) to 10 (impossible to perform an activity). The overall score is the mean of the 10 items and ranges from 0 to 10 with higher scores indicating more functional limitations. A negative change from Baseline in BASFI indicates improvement.
Change From Baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI) | Week 8,12,16,24
  The BASMI is a composite score based on 5 direct measurements of spinal mobility:
  cervical rotation (measured in degrees), tragus to wall distance (in centimeters [cm]) lumbar side flexion (in cm), lumbar flexion (modified Schober's) (in cm) and intermalleolar distance (in cm). Each measurement is converted to a linear score between 0 and 10. The total BASMI score is the average of the 5 scores and ranges from 0 to 10; the higher the BASMI score the more severe the patient's limitation of movement due to their ankylosing spondylitis. A negative change from Baseline indicates improvement.
Change From Baseline in Ankylosing Spondylitis Disease Activity Score (ASDAS) | Week 8,12,16,24
  ASDAS is a composite index to assess disease activity in Ankylosing Spondylitis. ASDAS combines the following 5 disease activity variables using a weighted formula:
  Patient's assessment of total back pain (BASDAI Question 2; NRS score 0 [none] - 10 [very severe]) Patient global assessment of disease activity (NRS score 0 [no activity] - 10 [severe activity]) Peripheral pain/swelling (BASDAI Question 3; NRS score 0 [none] - 10 [very severe]) Duration of morning stiffness (BASDAI Question 6; NRS score 0 [0 hours] - 10 [2 or more hours]) High-sensitivity C-reactive protein (hs-CRP) in mg/L. The overall score ranges from 0 with no defined upper score; published ranges for disease activity states as defined by the ASDAS include Inactive disease (ASDAS < 1.3) and very high disease (ASDAS > 3.5). A negative change from Baseline score indicates improvement in disease activity.
Change From Baseline in Ankylosing Spondylitis Quality of Life (ASQoL) Score | Week 8,12,16,24
  The ASQoL consists of 18 items related to quality of life, including the impact of pain on sleep, mood, motivation, ability to cope, activities of daily living, independence, relationships, and social life. Each item is answered as yes (scored as 1) or no (scored as 0).
  Scores are summed to obtain the overall score which ranges from 0 to 18, where higher scores indicate a worse quality of life. A negative change from Baseline in ASQoL indicates improvement in quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zeng, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China